CLINICAL TRIAL: NCT05136261
Title: A Pilot Study to Evaluate the Efficacy and Tolerability of Ceradan Advanced Moisturising Skin Barrier Cream in the Treatment of Children and Adolescents With Moderate Atopic Dermatitis
Brief Title: Evaluating the Efficacy and Tolerability of Ceradan Advanced Cream in the Treatment of Children With Atopic Dermatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYP2021/001
Record Dates: First submitted 2021-10-24; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Emollients will be dispensed in identical, unmarked containers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Ceradan Advanced Moisturising Skin Barrier cream - applied twice a day
  Interventions: Device: Ceradan ® Advanced Cream
- Control (Placebo Comparator): Aqueous Cream - applied twice a day
  Interventions: Device: Basic cream

INTERVENTIONS:
Device: Ceradan ® Advanced Cream — Ceradan ® Advanced Cream
  Arms: Treatment
Device: Basic cream — Basic cream
  Arms: Control

SUMMARY:
Atopic dermatitis is the most common chronic inflammatory skin condition worldwide and in Singapore. There is a significant impact on the quality of life as well as psychosocial burden on the patient and family. Emollients are one of the cornerstones in the treatment of atopic dermatitis and are frequently prescribed with topical anti-inflammatories such as topical corticosteroids or topical calcineurin inhibitors to be used during active flares. Emollients that have additional anti-inflammatory properties may be able to reduce usage of topical corticosteroids or calcineurin inhibitors. In this study the investigators hope to evaluate the use of a patented ceramide dominant emollient which sustainably lowers the skin pH (Ceradan ® Advanced Cream, Hyphens Pharma, Singapore) with a commonly prescribed emollient in Singapore (Basic Aqua Cream, ICM Pharma, Singapore) for the treatment of moderate atopic dermatitis in children and adolescents.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, controlled study comparing a patented ceramide dominant emollient which sustainably lowers the skin pH with a standard commercial emollient for the treatment of moderate atopic dermatitis over two weeks. Subjects will be concomitantly treated with a low-potency topical steroid (Desonide lotion, Galderma, France) at the start of the trial to minimize any underlying skin inflammation for a more comparable baseline skin state.

Investigators and subjects are blinded to the treatment allocation. Subjects will be randomized using a random number sequence in a 1:1 ratio between the two arms. The study administrator will keep this information concealed in an opaque, sealed envelope to be disclosed upon completion of the trial. Allocation is secure and concealed with no further changes to be made.

Subjects will be dispensed a mild potency topical steroid (Desonide lotion, Galderma, France) and 480g of emollient (Ceradan ® Advanced Cream, Hyphens Pharma, Singapore or Basic Cream, ICM Pharma, Singapore) for the duration of the trial. The amount of steroid dispense would depend on the weight of the subject (<20kg: 1 bottle, 20-40kg: 2 bottles, >40kg: 3 bottles). Emollients will be dispensed in identical, unmarked containers.

Subjects should not wash the test areas with water or cleansing products (e.g. soap, body cleansers, and bath and shower products) within the 12 hours prior to scheduled visit at 2 weeks (visit 1) for assessment. Subjects will be instructed to use mild potency topical steroid (Desonide lotion, Galderma, France), twice a day to all affected areas with eczema for the first three days of the trial. The topical steroid supplied can be used after the initial period of treatment as needed and subjects will be asked to record down the areas that treated and the duration of treatment. Subjects will be asked to use the emollient provided twice a day on the face, trunk, and limbs. This is to be used after application of topical steroids, where applicable. Subjects will be asked to not apply any other topical leave-on products (e.g. creams, lotions, ointments) on the test areas, apart from those products dispensed for this trial during the entire duration of the study. Subjects will be asked to apply the emollient on the test areas the last time within 3-12 hours before the scheduled final visit (visit 1). Dispensed product will be weighed and recorded prior to the start of the trial and on completion of the trial to assess the compliance and amount of product used.

Schedule of Visits

Assessment at baseline (Visit 0) includes:

* Baseline demographics (age, race and gender)
* Past medical history and drug allergies
* Family and personal history of atopy
* Atopic dermatitis history (duration of illness, areas affected, treatments used including type, frequency of use and amount of steroids/emollients used 1 month before enrollment)
* EASI score
* SCORAD score
* Skin pH (HI99181 pH Meter for Skin, Hanna Instruments Inc., Singapore)
* Transepidermal water loss (TEWL) (Delfin Technologies)
* Stratum corneum (SC) hydration (Delfin Technologies)
* Peak pruritus NRS (numerical rating scale) score
* Patient-Oriented Eczema Measure (POEM) score
* Patient Eczema Severity Time (PEST) score [11] via iControl Eczema Application (Hyphens Pharma, Singapore)
* Children's Dermatology Quality of Life (C-DLQI) score
* Teenagers' Quality of Life (T-QoL©) score
* Dermatitis Family Impact (DFI) Questionnaire

Assessment after 2 weeks (Visit 1) includes:

* EASI (Eczema Area and Severity Index) score
* SCORAD (Severity Scoring of Atopic Dermatitis) score
* Skin pH (HI99181 pH Meter for Skin, Hanna Instruments Inc., Singapore)
* TEWL (Delfin Technologies)
* SC hydration (Delfin Technologies)
* Peak pruritus NRS (numerical rating scale) score
* Patient-Oriented Eczema Measure (POEM) score
* Patient Eczema Severity Time (PEST) score via iControl Eczema Application (Hyphens Pharma, Singapore)
* Children's Dermatology Quality of Life (C-DLQI) score
* Teenagers' Quality of Life (T-QoL©) score
* Dermatitis Family Impact (DFI) Questionnaire

In the event of a severe exacerbation of atopic dermatitis, Visit 1 will be brought forward to allow the patient to return for an assessment and any rescue or additional treatment as required. The assessment measures planned after 2 weeks will be done at this visit as well.

Data Collection Methods Personal data will be treated as strictly confidential. Data will be collected using a secured encrypted database and anonymized. Data will be collected at baseline visit and follow up visit 2 weeks later. Further clarification will be made to the patient and/or family over phone call if required.

Potential difficulties and risks

* Adverse reactions and/or contact dermatitis to emollients or its constituents
* Burning or stinging sensation
* Increased itch
* Localized skin infections
* Exacerbation of atopic dermatitis
* Slips and falls

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged three to 16 years of age.
* Atopic dermatitis, in accordance with the U.K Working Party's Diagnostic Criteria.
* Moderate severity on both Eczema Area and Severity Index (EASI) and Scoring Atopic Dermatitis (SCORAD) scores. (I.e. 7.1-21 EASI and 29-48.9 SCORAD)
* Not currently infected eczema.
* Able to give informed consent or have a parent/guardian able and willing to give informed consent.

Exclusion Criteria:

* Known sensitivity or contact dermatitis to emollients, topical corticosteroids or any of its constituents.
* Currently infected eczema or frequent episodes of infected eczema requiring antibiotics.
* Currently on phototherapy, oral immunosuppressant, monoclonal antibodies for the treatment of eczema one month prior to start of study.
* Usage of any topical steroids or calcineurin inhibitors one week prior to start of study.
* Unable to give informed consent or have a parent/guarding unwilling to give consent.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in eczema severity and symptoms as determined by Eczema Area and Severity Index Score (EASI) | 2 weeks
  0=clear; 0.1-1=almost clear; 1.1-7=mild; 7.1-21=moderate; 21.1-50=severe; 50.1-72=very severe
Improvement in eczema severity and symptoms as determined by Severity Scoring of Atopic Dermatitis score (SCORAD) | 2 weeks
  The SCORAD score range is between 0 and 103 points and defines three classes of AD severity (i.e. mild if SCORAD <25, moderate if 25 ≤ SCORAD ≤ 50 and severe if SCORAD > 50)

SECONDARY OUTCOMES:
Changes in skin pH | 2 weeks
  Changes in skin pH will be measured with a pH meter - a lower pH value is desirable as the intervention is proposed to lower skin pH and help improve eczema
Changes in skin transepidermal water loss (TEWL) using a TEWL meter | 2 weeks
  A reduction in the amount of skin TEWL is desirable and expected for this trial
Changes in skin stratum corneum hydration | 2 weeks
  An increase in skin stratum corneum hydration is desirable and expected for this trial
Changes in POEM (Patient Oriented Eczema Measures) score | 2 weeks
  0-2 = clear/almost clear, 3-7 = mild, 8-16 = moderate, 17-24 = severe, and 25-28
Changes in PEST (Patient Eczema Severity Time) score | 2 weeks
  PEST is a picture-based score with 5 images associated with caregiver/patient-reported global severity assessment ranging from 1 ("not at all unhappy") to 5 ("extremely unhappy")
Changes in peak pruritus NRS (numerical response scale) scores | 2 weeks
  Peak Pruritus NRS score rates itch on a scale of 0-10 where 0 is no itch and 10 is the worst itch imaginable
Changes in C-DLQI (Children's Dermatology Quality of Life Index) scores | 2 weeks
  The C-DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired
Changes in T-QoL© scores | 2 weeks
  The T-QoL total score is calculated by summing the score of each of the 18 questions, resulting in a maximum of 36 and a minimum of 0.
  The questions in the T-QoL are divided into three parts (domains):
  Self-image (8 questions) Physical well-being and future aspirations (4 questions) Psychological impact and relationships (6 questions)
  The T-QoL score can also be reported as three separate scores:
  T-QoL self-image (score range 0-16) T-QoL physical/future (score range 0-8) T-QoL psychological/relationships (score range 0-12)
Changes in DFI scores | 2 weeks
  The minimum DFI score is 0 (= no impact on life of family). The maximum DFI score is 30 (= maximum effect on life of family).

OTHER OUTCOMES:
Adverse reactions | 2 weeks
  Adverse reactions experienced by subjects in the trial will be recorded
Amount of topical steroids used | 2 weeks
  Amount of topicals steroids used will be weighed pre and post trial

IPD SHARING:
Plan to Share IPD: Undecided